CLINICAL TRIAL: NCT03171844
Title: Early Skin to Skin in Neonatal reanimation_Risk Assessment in the Newborn With an Umbilical Venous Catheter
Brief Title: Early Skin to Skin in Neonatal Reanimation
Acronym: PA2PRéaNice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-AOI-01
Record Dates: First submitted 2017-05-29; First posted 2017-05-31 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Infant, Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin to skin (Experimental): Implement of skin to skin
  Interventions: Other: Skin to skin

INTERVENTIONS:
Other: Skin to skin — 3 sessions of skin to skin will be made on newborn wearing an umbilical venous catheter

SUMMARY:
In the reanimation neonatal department of the Nice's hospital, 34% of newborns admitted have an umbilical vein catheter (KTVO). Their parents are admitted 24h/24h by their side, where everything is done to set up the Attachment (participation in care, skin to skin, support of breastfeeding, ...).

The benefits of skin to skin described in developmental care of the newborn in the neonatal health services are well established. Nevertheless, for supposed risks (infectious and displacement of the catheter), registered in the memory of the teams, this care is not currently carried out when the newborns are carrying an umbilical venous catheter.

Sometimes, because of the presence of an umbilical venous catheter, parents and their newborns could not enjoy this moment of well-being in the first days of life. We therefore propose a study evaluating the current risks of skin to skin with an umbilical venous catheter by reflecting on a new protocol for laying and fixing this medical device.

ELIGIBILITY:
Inclusion Criteria:

* Newborn of gestational age less than 37SA
* Admitted in neonatal reanimation department at Nice's hospital
* Born in the maternity ward of the Nice's hospital
* Carriers of an umbilical venous catheter.

Exclusion Criteria:

* All newborns with medical contraindications from skin to skin:

  * Controlled hypothermia protocol
  * Newborn under HFO (High Frequency Oscillation)
  * Carrying a diaphragmatic hernia
  * Thoracic drain holder
  * With major PAH (hypertensive pulmonary artery)
* Symptomatic mother of acute infectious disease
* Mother whose physical or psychiatric capacity is not compatible with travel to the neonatal reanimation service within 3 days of delivery.
* Minor mother

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Bacteremia | 48h
  Occurrence of a bacterial blood infection concomitant with Umbilical venous catheter and up to 48 hours after its withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Florence CASAGRANDE, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France